CLINICAL TRIAL: NCT00226941
Title: A Phase 1-2 Trial of Cetuximab in Combination With Oxaliplatin, Capecitabine, and Radiation Therapy Followed by Surgical Resection for Locally-Advanced Rectal Cancer
Brief Title: A Phase 1-2 Trial of Cetuximab in Combination With Oxaliplatin, Capecitabine, and Radiation Therapy Followed by Surgery for Locally-advanced Rectal Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The response rate observed in the phase 1 portion of the study did not merit further evaluation in phase 2 portion of the study.
Sponsor: George Albert Fisher (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, George Albert Fisher, Professor of Medicine and Colleen Haas Chair in the School of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-12426; COR0001 (Other: OnCore); 95054 (Other: Stanford IRB, historical)
Record Dates: First submitted 2005-09-08; First posted 2005-09-27 (Estimated); Results first posted 2017-12-08 (Actual); Last update posted 2017-12-08 (Actual); Status verified 2017-11

CONDITIONS: Rectal Cancer; Colo-rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms; Colonic Neoplasms | interventions — Cetuximab; Oxaliplatin; Capecitabine; Radiotherapy; Diphenhydramine; Doxylamine

STUDY DESIGN:
Intervention Model Description: Sequential design for 4 dose combinations (arms) through phase 1
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 (Experimental): * Cetuximab 250 mg/m² / week
  * Capecitabine 800 mg/m²
  * Radiotherapy (XRT)
  * Oxaliplatin 100 mg/m², Days 2 and 23
  Interventions: Drug: Cetuximab; Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Radiotherapy; Drug: Diphenhydramine hydrochloride (HCl)
- Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 (Experimental): * Cetuximab 250 mg/m² / week
  * Capecitabine 700 mg/m²
  * Radiotherapy (XRT)
  * Oxaliplatin 85 mg/m², Days 2 and 23
  Interventions: Drug: Cetuximab; Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Radiotherapy; Drug: Diphenhydramine hydrochloride (HCl)
- Group A - Cetuximab + Capecitabine-800 + XRT (Experimental): * Cetuximab 250 mg/m² / week
  * Capecitabine 800 mg/m²
  * Radiotherapy (XRT)
  Interventions: Drug: Cetuximab; Drug: Capecitabine; Radiation: Radiotherapy; Drug: Diphenhydramine hydrochloride (HCl)
- Group B - Cetuximab + Capecitabine-1000 + XRT (Experimental): * Cetuximab 250 mg/m² / week
  * Capecitabine 1000 mg/m²
  * Radiotherapy (XRT)
  Interventions: Drug: Cetuximab; Drug: Capecitabine; Radiation: Radiotherapy; Drug: Diphenhydramine hydrochloride (HCl)

INTERVENTIONS:
Drug: Cetuximab — Cetuximab is a chimeric anti-epidermal growth factor receptor (anti-EGFR) monoclonal antibody, administered via a intravenous (IV) infusion at 400 mg/m² (initial loading dose) or 250 mg/m² (weekly dose). Dosage is based on m² of body surface area (BSA)
  Other Names: Erbitux; C225; IMC-C225
Drug: Oxaliplatin — Oxaliplatin is a cancer medication used to treat colorectal cancer, and is administered on Days 2 and 23.
  Other Names: Eloxatin
  Arms: Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100; Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85
Drug: Capecitabine — Capecitabine is a cancer medication, and is administered based on m² of body surface area (BSA) delivered in equivalent morning and evening doses
  Other Names: Xeloda
Radiation: Radiotherapy — Radiotherapy is administered on weekdays in 180 centigray fractions ("doses"), for 28 total fractions delivering a total dose of 5040 centigray (cGy)
  Other Names: XRT
Drug: Diphenhydramine hydrochloride (HCl) — Diphenhydramine HCl 50 mg (or equivalent) is administered as a per-medication for cetuximab
  Other Names: Benadryl; Unisom; Sominex

SUMMARY:
The objectives of this study are to:

1. To assess dose-limiting toxicities (DLTs) of capecitabine +/- oxaliplatin in a combination regimen with capecitabine and radiotherapy (Phase 1)
2. To determine the maximum-tolerated dose (MTD) when capecitabine

   * oxaliplatin in a combination regimen with capecitabine and radiotherapy (Phase 1)
3. To determine the pathologic response rate of cetuximab +/- oxaliplatin in combination with capecitabine and radiotherapy (Phase 2)

DETAILED DESCRIPTION:
Part of the treatment plan for this study is surgical removal of the tumor that is planned to occur 6 to 8 weeks after completion of radiotherapy (XRT). This study consists of 2 distinct phases (Phase 1 and Phase 2).

In Phase 1, the objectives are to

1. Assess dose-limiting toxicities (DLTs) and
2. Determine a maximum-tolerated dose (MTD)

The Phase 1 endpoints are assessed on an initial cohort of patients after the completion of the chemo-radiotherapy regimen at defined timepoints that precede surgery.

Phase 2 is the efficacy assessment portion of this study. In Phase 2, the objective is to accrue an expansion cohort. Efficacy assessments for phase 2 are to be assessed across all study participants at the time of, or after, surgery, as measured by the pathologic response rate; downstaging; and survival at 5 years from the start of treatment.

ELIGIBILITY:
INCLUSION CRITERIA

* Histologically-confirmed adenocarcinoma of the rectum. Clinical stages T3; T4; or N1 as determined by endoscopic ultrasound; or a rectal CT or MRI scan are eligible, including T3 N0; T3 N1; T4 N0; T4 N1; T1-4 N1. Rectal cancers are defined as those whose distal border extends to within 12 cm of the anal verge.
* Age ≥ 18
* Karnofsky performance status (KPS) ≥ 70
* Leukocyte count > 3,500 x 10e6/µL
* Platelet count > 100,000/µL
* Serum glutamic-oxaloacetic transaminase (SGOT) < 2.5 x institutional upper limits of normal (ULN)
* Serum glutamic-pyruvic transaminase (SGPT) < 2.5 x ULN
* Alkaline phosphatase < 2.5 x ULN
* Total bilirubin < 1.5x ULN
* Creatinine:

  * Within normal institutional limits
  * OR
  * Creatinine clearance > 60 mL/min/1.73 m2 (if serum creatinine levels above institutional normal)
* Ability to swallow pills without difficulty
* Women of child-bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG), within 72 hours prior to the start of study medication
* Women of child-bearing potential must be using an adequate method of contraception to avoid pregnancy throughout the treatment

EXCLUSION CRITERIA

* Metastatic (M1) or stage IV disease
* Prior history of treatment with cetuximab or other therapy targeting EGFR
* Prior history of anti-cancer murine monoclonal antibody therapy
* Prior pelvic or whole abdominal radiotherapy
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness / social situations that would limit compliance with study requirements
* Patients with a concurrent malignancy or previous malignancy within 5 years of screening will be excluded from this study (EXCEPTION: concurrent or previous non-melanoma skin cancer, hematolymphoid malignancy or carcinoma in-situ of the cervix may be allowed at the investigator's discretion)
* Inability to sign written consent
* Pregnant or breastfeeding
* Unwilling or unable to use effective contraception in self or partner for the entire study period and for up to 4 weeks after the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-06; Primary Completion 2008-03 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George A Fisher, MD, PhD, Principal Investigator — Stanford University; Branimir I Sikic, MD, Study Chair — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85: * Cetuximab 250 mg/m² / week
  * Capecitabine 700 mg/m²
  * Radiotherapy (XRT)
  * Oxaliplatin 85mg/m², Days 2 and 23
- Group A - Cetuximab + Capecitabine-800 + XRT; Group B - Cetuximab + Capecitabine-1000 + XRT: * Cetuximab 250 mg/m² / week
  * Capecitabine 1000 mg/m²
  * Radiotherapy (XRT)
Period: Overall Study
Arm/Group | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 | Group A - Cetuximab + Capecitabine-800 + XRT | Group B - Cetuximab + Capecitabine-1000 + XRT
Started | 6 | 6 | 4 | 7
Completed | 6 | 6 | 4 | 5
Not Completed | 0 | 0 | 0 | 2
Not completed — Withdrawal by subject - toxicity | 0 | 0 | 0 | 1
Not completed — Withdrawn by investigator - unrelated AE | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 | Group A - Cetuximab + Capecitabine-800 + XRT | Group B - Cetuximab + Capecitabine-1000 + XRT | Total
Number analyzed (Participants) | 6 | 6 | 4 | 7 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 4 | 5 | 20
  >=65 years | 1 | 0 | 0 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 2 | 5
  Male | 5 | 4 | 4 | 5 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 6 | 4 | 6 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 4 | 6 | 4 | 5 | 19
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Histology [Count of Participants; unit: Participants]
  Adenocarcinoid Tumor | 0 | 0 | 1 | 4 | 5
  Adenocarcinoma, Nos | 6 | 6 | 2 | 3 | 17
  Adenosarcoma | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity (DLT) - Number of DLTs by Treatment Group
Description: Dose-limiting Toxicity (DLT) is the measure used to establish overall Maximum-tolerated dose (MTD) of cetuximab + capecitabine + radiotherapy +/- oxaliplatin. MTD is defined as the highest dose level for which participants have a < 30% incidence of dose-limiting toxicity (DLT). The outcome is expressed as the number of DLTs by treatment group.
Time Frame: 10 weeks
Population: All participants were formally part of the phase 1 portion of this study.
Measure: Number; unit: DLTs
Arm/Group | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 | Group A - Cetuximab + Capecitabine-800 + XRT | Group B - Cetuximab + Capecitabine-1000 + XRT
Number analyzed (Participants) | 6 | 6 | 4 | 7
DLTs | 10 | 2 | 0 | 0

2. Primary Outcome: Dose-limiting Toxicity (DLT) - Number of Participants Affected
Description: Dose-limiting Toxicity (DLT) is the measure used to establish overall Maximum-tolerated dose (MTD) of cetuximab + capecitabine + radiotherapy +/- oxaliplatin. MTD is defined as the highest dose level for which participants have a < 30% incidence of dose-limiting toxicity (DLT). The outcome is expressed as the number of participants experiencing a DLT.
Time Frame: 10 weeks
Population: All participants were formally part of the phase 1 portion of this study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 | Group A - Cetuximab + Capecitabine-800 + XRT | Group B - Cetuximab + Capecitabine-1000 + XRT
Number analyzed (Participants) | 6 | 6 | 4 | 7
Participants | 4 | 2 | 0 | 0

3. Secondary Outcome: Pathologic Response Rate
Description: After treatment with capecitabine, cetuximab, radiotherapy, and oxaliplatin, the pathologic response rate was assessed based on the excised tumor taken at the time of surgical resection. Pathologic response rate was determined as the number and proportion of participants who experienced either downstaging of their disease, or complete response (CR, no detectable disease). A participant will be considered to have downstaging of the tumor as a result of the neoadjuvant therapy when the primary tumor (T) stage by pathology isless than the T stage by clinical (endoscopic) evaluation, or when the regional lymph node (N) tumor stage by pathology is less than the N stage by clinical (endoscopic) evaluation.
Time Frame: 12 to 14 weeks after radiotherapy
Population: This outcome is specifically defined per protocol as the phase 2 portion of the study, which did not occur. However, the data for this measure are available from the phase 1 participants (only), and are provided for completeness.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 | Group A - Cetuximab + Capecitabine-800 + XRT | Group B - Cetuximab + Capecitabine-1000 + XRT
Number analyzed (Participants) | 5 | 6 | 4 | 5
Participants | 4 | 5 | 3 | 5

4. Secondary Outcome: Tumor Downstaging at Surgical Resection
Description: Downstaging means a reduction from the stage of disease observed at baseline to the stage of disease after treatment with cetuximab, radiotherapy, oxaliplatin, and capecitabine, as determined at the time of surgical removal of the tumor. Downstaging may be observed as improvements in tumor staging at the primary site of the tumor; in nearby (regional) lymph nodes; or in metastatic disease beyond the regional lymph nodes. This outcome specifically does not include participants that achieved a complete response, nor those that experienced no response or disease progression.
Time Frame: 12 to 14 weeks after radiotherapy
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100; Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85: * Cetuximab 250 mg/m² / week
  * Capecitabine 700 mg/m²
  * Radiotherapy (XRT)
  * Oxaliplatin 85 mg/m², Days 2 and 23
Arm/Group | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 | Group A - Cetuximab + Capecitabine-800 + XRT | Group B - Cetuximab + Capecitabine-1000 + XRT
Number analyzed (Participants) | 5 | 6 | 4 | 5
Participants | 4 | 5 | 3 | 5

5. Secondary Outcome: Time-to-Progression (TTP)
Description: Time-to-progression was assessed as the time from the date of surgical resection to the appearance of either local disease recurrence or distant metastases by any modality (eg, clinical exam, endoscopy, radiographic imaging). All relapses were to be confirmed by biopsy and pathology review.
Time Frame: 5 years
Population: This study was terminated before all patients reached 5 years from the date of surgical resection. Only patients that progressed are reported, and since no patients progressed in Group 2, median and range are not reportable.
Measure: Median (Full Range); unit: years
Groups:
- Group 2 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-85: * Cetuximab 250 mg/m² / week
  * Capecitabine 700 mg/m²
  * Radiotherapy (XRT)
  * Oxaliplatin 85 mg/m², Days 2 and 23
Arm/Group | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 | Group 2 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-85 | Group A - Cetuximab + Capecitabine-800 + XRT | Group B - Cetuximab + Capecitabine-1000 + XRT
Number analyzed (Participants) | 2 | 0 | 1 | 3
years | 1.4 [0.8 to 2.0] |  | 3.0 [3.0 to 3.0] | 3.9 [0.2 to 5.0]

6. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was assessed as the mean survival from the date of entry on study though 72 months.
Time Frame: 72 months
Population: This outcome is defined per protocol as study phase 2, which did not occur. However, data are provided for phase 1 participants, for completeness. This study was terminated before all patients reached 5 years on study. Some patients are reported as the last known alive date.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 | Group A - Cetuximab + Capecitabine-800 + XRT | Group B - Cetuximab + Capecitabine-1000 + XRT
Number analyzed (Participants) | 6 | 6 | 4 | 5
months | 59.7 (0.7) | 57.0 (5.8) | 54.4 (11.1) | 53.7 (11.3)

7. Secondary Outcome: Survival at 5 Years
Description: Survival at 5 years was assessed as the number of participants alive 5 years after starting treatment.
Time Frame: 5 years
Population: This outcome is defined per protocol as study phase 2, which did not occur. However, data are available from the phase 1 participants (only), and are provided for completeness. This study was terminated before all patients reached 5 years from study entry. Only patients known to be alive at 5 years are reported.
Measure: Count of Participants; unit: Participants
Groups:
- Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85: * Cetuximab 250 mg/m² / week
  * Capecitabine 700 mg/m²
  * Radiotherapy (XRT)
  * Oxaliplatin 850 mg/m², Days 2 and 23
- Group B - Cetuximab + Capecitabine-800 + XRT: * Cetuximab 250 mg/m² / week
  * Capecitabine 1000 mg/m²
  * Radiotherapy (XRT)
Arm/Group | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 | Group A - Cetuximab + Capecitabine-800 + XRT | Group B - Cetuximab + Capecitabine-800 + XRT
Number analyzed (Participants) | 6 | 6 | 4 | 5
Participants | 5 | 4 | 3 | 3

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 | Group A - Cetuximab + Capecitabine-800 + XRT | Group B - Cetuximab + Capecitabine-1000 + XRT
All-Cause Mortality (participants affected / at risk) | 1/6 | 1/6 | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 3/4 | 7/7
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 4/4 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 (N=6) | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 (N=6) | Group A - Cetuximab + Capecitabine-800 + XRT (N=4) | Group B - Cetuximab + Capecitabine-1000 + XRT (N=7)
Decrease in lung volumes with increased bibasilar atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Small bowel obstruction-Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 3 (4) | 1 (1) | 2 (2) | 1 (1)
Dehydration (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (8) | 2 (7) | 0 (0) | 5 (12)
Nausea (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 1 (2) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 - Cetuximab + Capecitabine-800 + XRT + Oxaliplatin-100 (N=6) | Group 2 - Cetuximab + Capecitabine-700 + XRT + Oxaliplatin-85 (N=6) | Group A - Cetuximab + Capecitabine-800 + XRT (N=4) | Group B - Cetuximab + Capecitabine-1000 + XRT (N=7)
Abdominal cramping (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 4 (4) | 1 (1) | 3 (3) | 2 (2)
Pain (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Libido (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Dry eye syndrome (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Edema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (Immune system disorders) | 4 (7) | 1 (2) | 2 (2) | 1 (1)
Insomnia (Investigations) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Rigors (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Fever (Infections and infestations) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Hemorrhage in rectum (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Syncope (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Depression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Backache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bilateral jaw pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Distension (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Bloody stool (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 4 (5)
Bloody rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body aches (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Candidal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Chest tightness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cold sensitivity (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (2) | 1 (1) | 0 (0)
Constipation, alternating with diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Skin cracking (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (2) | 0 (0) | 3 (3)
Cramping (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Cuticle dryness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dehydration (General disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (10) | 2 (7) | 0 (0) | 4 (11)
Diarrhea with cramping (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated alanine aminotransferase (ALT) (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Elevated aspartate aminotransferase (AST) (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema at incision (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatus (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Flu-like symptoms (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flushing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash, follicular, chest and back (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain, groin (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hand and foot syndrome (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypomagnesemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Left arm numbness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain, left knee (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lightheadedness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abnormal liver function test (LFT) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain, lower back (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low grade fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hematocrit decreased (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 6 (14) | 1 (2) | 2 (2) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain with bowel movements (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (2) | 3 (3)
Weight loss (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (4) | 2 (2) | 0 (0) | 1 (1)
Infection, urinary track (UTI) (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitancy (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection, upper respiratory tract (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0
Pain, umbilical cord protrusion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tingling, fingertips (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tingling, cheeks (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Taste disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Skin dryness (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood in stool, scant (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy, right arm (Nervous system disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Reflux (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection, rectal-anal (General disorders) | 3 (3) | 5 (6) | 2 (2) | 2 (2)
Radiation demititis (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (11) | 6 (10) | 4 (7) | 5 (12)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 2 (2) | 4 (5) | 1 (1) | 2 (2)
Pain (t11-12 level) (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain, bladder and testes (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain, middle ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain, throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial was halted after the phase 1 portion of enrollment, and before the phase 2 portion accrued.

Data reported for phase 2 objectives/outcomes do not include any phase 2 participants, and are only provided for completeness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No